CLINICAL TRIAL: NCT07375069
Title: Characterization of Cardiovascular Risk Profile and Therapeutic Management in Patients With Type 2 Diabetes Mellitus in Italy - CardioMET Registry
Brief Title: Characterization of Cardiovascular Risk Profile and Therapeutic Management in Patients With Type 2 Diabetes Mellitus in Italy
Acronym: CardioMET
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Pasquale Perrone Filardi, Professor, Federico II University
Other Study IDs: Prot. 189/2022
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data collection — Data collection on diabetes therapy and follow-up

SUMMARY:
CardioMET is an observational, multicenter, real-life registry, intending to collect data on patients with Type 2 Diabetes Mellitus, attending internal medicine and cardiology outpatient clinics. The aim of the registry is to characterize the cardiovascular risk profile and pharmacological management of Type 2 Diabetes Mellitus in Italy, in accordance with current ESC and AHA guidelines for primary and secondary prevention of CV disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Diagnosis of type 2 diabetes mellitus (T2DM);
* Ability to understand the study procedures and provide written informed consent.

Exclusion Criteria:

* Known or suspected liver disease;
* Patients with type 1 diabetes mellitus;
* Cardiac surgery or percutaneous coronary revascularization scheduled within the next 3 months;
* Patients with acute inflammatory or infectious diseases during the previous 3 months;
* Patients with chronic inflammatory, immune, or infectious diseases;
* Patients with ongoing malignant neoplasms;
* History of alcohol, drug, or medication abuse;
* Clinically significant hematological disorders;
* Systemic steroid treatment within the last 6 months;
* Acute-phase metabolic disorders;
* Any condition that may put the patient at risk by participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive diabetic patients attending the outpatient clinics, in primary and secondary prevention of cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Diabetes treatment adherence according to the most recent European Guidelines | 12-24-36-48 months
  Outpatients clinic treatment adherence will be measured as the percentage of patients receiving guideline-directed medical therapy prescriptions.

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University of Naples, Department of Advanced Biomedical Sciences, Napoli, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No